CLINICAL TRIAL: NCT00462189
Title: A Phase 1, Multicenter, Dose Escalation Study of CAT-8015 in Patient With Relapsed or Refractory Hairy Cell Leukemia (HCL)
Brief Title: Safety Study of CAT-8015 Immunooxin in Patients With HCL With Advance Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge Antibody Technology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1001
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Leukemia; Hairy Cell Leukemia; HCL
Keywords: CAT-8015; HA22; HCL; Relapse; Refractory; immunotherapy; immunotoxin
MeSH Terms: conditions — Leukemia; Leukemia, Hairy Cell; Recurrence | interventions — immunotoxin HA22; Biological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Immunotoxin therapy
Drug: CAT-8015 Immunotoxin
Procedure: Biological therapy

SUMMARY:
RATIONALE: The CAT-8015 immunotoxin can bind tumor cells and kill them without harming normal cells. This may be an effective treatment for hairy cell leukemia(HCL) that has not responded to chemotherapy, surgery or radiation therapy.

PURPOSE: Phase I dose escalation study to determine the maximum tolerated dose of CAT-8015 immunotoxin in treating patients who have hairy cell leukemia (HCL) that has not responded to treatment.

DETAILED DESCRIPTION:
OUTLINE: Patients receive CAT-8015 IV over 30 minutes on days 1, 3, and 5 followed by rest. Treatment repeats every 4 weeks for up to a total of 10 courses in the absence of dose limiting toxicity, complete response or disease progression. Patients are followed at 1, 3, 6,12,15,18, 21, 24 months following the start of the last treatment cycle.

Cohorts of 3-6 patients each will receive escalating doses of recombinant CAT-8015 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose proceeding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, between16 to 25 new patients will be added to the MTD cohort depending on how well the CAT-8015 is tolerated.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS:

* Confirmed diagnosis of hairy cell leukemia
* Measurable disease

At least one of the following indications for treatment:

* Neutropenia (ANC <1000 cells/µL)
* Anemia (Hgb <10g/dL)
* Thrombocytopenia (Plt <100,000/µL)
* An absolute lymphocyte count of >20,000 cells/µL, or
* Symptomatic splenomegaly
* Patient's must have had at least 2 prior systemic therapies. There must have been at least 2 prior courses of purine analog, or 1 if the response to this course lasted <2 years, or if the patient had unacceptable toxicity to purine analog.

PATIENT CHARACTERISTICS:

Performance status • ECOG 0-2

Life expectancy

• Life expectancy of greater than 6 months, as assessed by the principal investigator

Other

* Patients with other cancers who meet eligibility criteria and have had less than 5 years of disease free survival will be considered on a case-by-case basis
* Ability to understand and sign informed consent
* Female and male patients agree to use an approved method of contraception during the study

EXCLUSION CRITERIA:

* Documented and ongoing central nervous system involvement with their malignant disease (history of CNS involvement is not an exclusion criterion)
* History of bone marrow transplant
* Pregnant or breast-feeding females
* Patients whose plasma contains either a significant level of antibody to CAT-8015 as measured by ELISA, or antibody that neutralizes the binding of CAT-8015 to CD22 as measured by a competition ELISA.
* HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs)
* Hepatitis B surface antigen positive
* Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements

Hepatic function: serum transaminases (either ALT or AST) or bilirubin:

• ≥ Grade 2, unless bilirubin is due to Gilbert's disease

Renal function: serum creatinine clearance ≤60mL/min as estimated by Cockroft-Gault formula

Hematologic function:

* The ANC <1000/cmm, or platelet count <50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy)
* Baseline coagulopathy > grade 3 unless due to anticoagulant therapy
* A patient will not be excluded because of pancytopenia ≥ Grade 3, or erythropoietin dependence, if it is due to disease, based on the results of bone marrow studies

Pulmonary function:

• Patients with < 50% of predicted forced expiratory volume (FEV1) or <50% of predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin concentration and alveolar volume. Note: Patients with no prior history of pulmonary illness are not required to have PFTs. FEV1 will be assessed following bronchodilator therapy.

Recent prior therapy:

* Cytotoxic chemotherapy (except stable doses of prednisone), whole body electron beam radiation therapy, interferon, retinoids or other systemic therapy, or investigational therapy of the malignancy for 3 weeks prior to entry into the trial
* Less than or equal to < 3 months prior monoclonal antibody therapy (i.e. rituximab)
* Patients who have received or are receiving radiation therapy less than 3 weeks prior to study entry will be not be excluded providing the volume of bone marrow treated is less than 10% and also the patient has measurable disease outside the radiation port
* Any history of pseudomonas-exotoxin (PE) immunotoxin administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-04

PRIMARY OUTCOMES:
Estimate the maximum dose that can be safely administered to a patient
Characterize the toxicity profile of CAT-8015
Study the clinical pharmacology of CAT-8015
Observe anti-tumor activity, if any.

SECONDARY OUTCOMES:
To assess the immunogenic potential of CAT-8015 to induce antibodies
To investigate the potential of biomarkers to predict any therapeutic or toxic response.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Cancer Center of Northwestern University, Chicago, Illinois
  - Warren Grant Megnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
- Klinika Hamtologii Uniwersytetu Medycznego (Medical University of Lodz), Lodz, Poland
- Royal Marsden Hospital and Institute of Cancer Research, Surrey, United Kingdom

REFERENCES:
- [Background] Kreitman RJ, Squires DR, Stetler-Stevenson M, Noel P, FitzGerald DJ, Wilson WH, Pastan I. Phase I trial of recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) in patients with B-cell malignancies. J Clin Oncol. 2005 Sep 20;23(27):6719-29. doi: 10.1200/JCO.2005.11.437. Epub 2005 Aug 1. PMID 16061911
- [Derived] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230